CLINICAL TRIAL: NCT05169047
Title: The Holistic Response of Patients With Persistent Spinal Pain Syndrome Type II by Subthreshold Spinal Cord Stimulation Compared to Best Medical Treatment, Investigated by a Multicentric Randomized Controlled Trial
Brief Title: Subthreshold SCS or BMT
Acronym: TRADITION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRADITION
Record Dates: First submitted 2021-11-29; First posted 2021-12-23 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Medical Treatment (Active Comparator)
  Interventions: Other: Best Medical Treatment
- Subthreshold Spinal Cord Stimulation (Active Comparator)
  Interventions: Other: Subthreshold Spinal Cord Stimulation

INTERVENTIONS:
Other: Best Medical Treatment — For each patient who is randomized to BMT, an optimal individual treatment plan will be developed by the treating physician.
  Arms: Best Medical Treatment
Other: Subthreshold Spinal Cord Stimulation — SCS will be programmed at subthreshold stimulation.
  Arms: Subthreshold Spinal Cord Stimulation

SUMMARY:
Given the substantial socioeconomic impact of Spinal Cord Stimulation (SCS) implantations and given that currently no direct high-quality evidence with a relevant outcome measurement is available to guide the treatment choice between subthreshold SCS versus best medical treatment in patients with Persistent Spinal Pain Syndrome Type 2 (PSPS-T2), we here propose a scientifically well-constructed randomized controlled trial to answer this question.

The primary scientific objective is to examine whether subthreshold SCS, compared to best medical treatment, provided to patients with PSPS-T2 results in a higher percentage of clinical holistic responders at 6 months. The secondary objective of the study is to examine if subthreshold SCS compared with BMT is having more efficacy in improving patients' individual competencies for self-management, increasing the likelihood to return to work, work status and healthcare expenditure, improving pain relief, obtaining pain medication reduction, decreasing anxiety and depression, increasing quality of life and decreasing disability.

DETAILED DESCRIPTION:
After filling in the questionnaires at the 6 months follow-up visit, patients could change treatment groups (in both directions). This decision will be a shared decisions between patient and treating physician in case the randomized intervention did not provided enough pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Persistent Spinal Pain Syndrome Type II (PSPS-T2)
* Chronic pain as a result of PSPS-T2 that exists for at least 6 months with a pain intensity of at least 4/10 on the Numeric Rating Scale, refractory to conservative treatment.
* PSPS-T2 patients eligible for subthreshold SCS
* Age > 18 years
* Patient has been informed of the study procedures and has given written informed consent
* Patient willing to comply with study protocol including attending the study visits

Exclusion Criteria:

* Expected inability of patients to receive or properly operate the spinal cord stimulation system
* Evidence of an active psychiatric disorder
* Suffering from another chronic illness characterised by chronic generalized widespread pain (e.g. rheumatoid arthritis, fibromyalgia, chronic fatigue syndrome, scleroderma).
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Clinical holistic responder status | The change between the baseline screening and the evaluation at 1 month, 6 months and 12 months.
  The clinical holistic responder status as a composite measure represents the global effect of a treatment, based on a combination of questionnaires.

SECONDARY OUTCOMES:
Overall pain intensity with Visual Analogue Scale (VAS) | The change between the baseline screening and the evaluation at 1 month, 6 months and 12 months.
  Overall pain, defined as a combination of back and leg pain, but not pain from other body parts, measured with the VAS (100mm)
Pain medication use | The change between the baseline screening and the evaluation at 1 month, 6 months and 12 months.
  Open question regarding the dosage, frequency and type of pain medication
Functional disability | The change between the baseline screening and the evaluation at 1 month, 6 months and 12 months.
  The functional disabilities will be assessed with the Oswestry Disability Index (ODI)
Health related quality of life | The change between the baseline screening and the evaluation at 1 month, 6 months and 12 months.
  Health related quality of life, evaluated with the EuroQol with five dimensions and 5 levels
Patient global impression of change | Evaluated at 1 month, 6 months and 12 months.
  Patients will be asked to quantify the impression of change after treatment using the Patient Global Impression of Change scale (PGIC).
Work status | The change between the baseline screening and the evaluation at 1 month, 6 months and 12 months.
  Work status is evaluated with a self-designed questionnaire
Patients' individual competencies for self-management | The change between the baseline screening and the evaluation at 1 month, 6 months and 12 months.
  Patient activation measure-13 (PAM) is a 13-item instrument which assesses self-reported behaviour, knowledge, and confidence for self-management of one's health.
Healthcare utilisation. | The change between the baseline screening and the evaluation at 1 month, 6 months and 12 months.
  Healthcare expenditure will be investigated by self-reporting methods.
Anxiety and Depression. | The change between the baseline screening and the evaluation at 1 month, 6 months and 12 months.
  The hospital Anxiety and Depression Scale (HADS) will measure symptoms of anxiety and depression

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (5):
  - Jessa Ziekenhuis, Hasselt
  - Universitair Ziekenhuis Brussel, Jette
  - Emmaüs, AZ Sint-Maarten, Mechelen
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout

REFERENCES:
- [Derived] Goudman L, Putman K, Van Doorslaer L, Billot M, Roulaud M, Rigoard P; TRADITION consortium; Moens M. Proportion of clinical holistic responders in patients with persistent spinal pain syndrome type II treated by subthreshold spinal cord stimulation compared to best medical treatment: a study protocol for a multicentric randomised controlled trial (TRADITION). Trials. 2023 Feb 20;24(1):120. doi: 10.1186/s13063-023-07140-3. PMID 36803412
- See also: Study protocol — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9940414/